CLINICAL TRIAL: NCT05578079
Title: The Effectiveness of Music on Pain During Heel Blood Collection in Premature Infants: A Double-Blind Randomized Controlled Trial
Brief Title: The Effectiveness of Music on Pain During Heel Blood Collection in Premature Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Pınar Dogan, Research Ass., Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 05
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Pain
Keywords: Premature; Pain; Music
MeSH Terms: conditions — Pain; Premature Birth | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No music will be played to the control group.
- Intervention 1 (Active Comparator): The Intervention-1 group will listen to the music which determined by the researchers by examining the literature (DOI: 10.4274/jpr.24892). The music which determined by the researchers is "The art of fugue" by Johann Sebastian Bach.
  Interventions: Other: Music
- Intervention 2 (Active Comparator): The Intervention-2 group will listen to lullaby.
  Interventions: Other: Music

INTERVENTIONS:
Other: Music — Intervention-1 group will listen to the classical music that the "Arts of Fugue" by Bach.
  Arms: Intervention 1
Other: Music — Intervention-2 group will listen to lullaby.
  Arms: Intervention 2

SUMMARY:
Premature babies receiving treatment and care in the Neonatal Intensive Care Unit (NICU) are exposed to various painful procedures. Repetitive and untreated painful procedures have a negative impact on the physiological, cognitive and behavioral development of the baby.

Various approaches such as white noise, music, lullaby, kangaroo care, breastfeeding, swaddling, massage, and therapeutic positioning are used to reduce the painful processes that newborns are exposed to in the NICU.

DETAILED DESCRIPTION:
Premature babies receiving treatment and care in the Neonatal Intensive Care Unit (NICU) are exposed to various painful procedures. Repetitive and untreated painful procedures have a negative impact on the physiological, cognitive and behavioral development of the baby.

Various approaches such as white noise, music, lullaby, kangaroo care, breastfeeding, swaddling, massage, and therapeutic positioning are used to reduce the painful processes that newborns are exposed to in the NICU.

ELIGIBILITY:
Inclusion Criteria:

* Parent being voluntary to participate in the study
* Being born at 32-36+6 gestastional week
* The baby's condition is stable
* Having passed hearing test
* Having not congenital malformation

Exclusion Criteria:

* Birth weight below 2500 g
* Receiving analgesics or sedatives
* Need for mechanical ventilation
* Heel blood collection is not successful in the first time

Ages: 32 Weeks to 37 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-10-14 (Actual); Primary Completion 2023-04-25 (Actual); Study Completion 2023-04-25 (Actual)

PRIMARY OUTCOMES:
Baby's heart rate | 2 minutes before collecting heel blood
  The baby's pulse rate will be measured.
Baby's heart rate | During heel blood collection
  The baby's pulse rate will be measured.
Baby's heart rate | 2 minutes after collecting heel blood
  The baby's pulse rate will be measured.
Baby's respiratory rate | 2 minutes before collecting heel blood
  The baby's respiratory rate will be measured.
Baby's respiratory rate | During heel blood collection
  The baby's respiratory rate will be measured.
Baby's respiratory rate | 2 minutes after collecting heel blood
  The baby's respiratory rate will be measured.
Baby's oxygen saturation | 2 minutes before collecting heel blood
  The baby's oxygen saturation will be measured.
Baby's oxygen saturation | During heel blood collection
  The baby's oxygen saturation will be measured.
Baby's oxygen saturation | 2 minutes after collecting heel blood
  The baby's oxygen saturation will be measured.
Premature Infant Pain Profile (PIPP) | 2 minutes before collecting heel blood
  PIPP scores will be evaluated separately by two experts in the field.
Premature Infant Pain Profile (PIPP) | During heel blood collection
  PIPP scores will be evaluated separately by two experts in the field.
Premature Infant Pain Profile (PIPP) | 2 minutes after collecting heel blood
  PIPP scores will be evaluated separately by two experts in the field.

CONTACTS AND LOCATIONS:
Overall Officials: Defne ENGUR, Assoc.Prof., Study Chair — Tepecik Research and Training Hospital
Locations (1):
- Tepecik Research and Training Hospital, Izmir, Turkey (Türkiye)